CLINICAL TRIAL: NCT04779177
Title: An Open-label Multiple Oral Dose Study to Determine the Safety, Tolerability, and Pharmacokinetics of Lumateperone in Patients, Ages 13 to 17 Years, Diagnosed With Schizophrenia or Schizoaffective Disorder
Brief Title: Safety, Tolerability, and Pharmacokinetics of Lumateperone in Pediatric Patients With Schizophrenia or Schizoaffective Disorder
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Intra-Cellular Therapies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ITI-007-020
Record Dates: First submitted 2021-02-26; First posted 2021-03-03 (Actual); Results first posted 2025-11-12 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-10

CONDITIONS: Schizophrenia; Pediatric
MeSH Terms: conditions — Schizophrenia | interventions — lumateperone

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lumateperone 42 mg once daily for 5 days (Experimental)
  Interventions: Drug: Lumateperone 42 mg
- Lumateperone 28 mg once daily for 5 days (Experimental)
  Interventions: Drug: Lumateperone 28 mg

INTERVENTIONS:
Drug: Lumateperone 42 mg — Lumateperone 42 mg, oral administration
  Arms: Lumateperone 42 mg once daily for 5 days
Drug: Lumateperone 28 mg — Lumateperone 28 mg, oral administration
  Arms: Lumateperone 28 mg once daily for 5 days

SUMMARY:
Study ITI-007-020 is a Phase 1b, multicenter, open-label study to evaluate the safety, tolerability, and PK of lumateperone as treatment for adolescent patients with schizophrenia or schizoaffective disorder.

ELIGIBILITY:
Main Inclusion Criteria:

* Male or female patients between 13 and 17 years of age, inclusive
* Clinical diagnosis of schizophrenia or schizoaffective disorder according to Diagnostic and Statistical Manual of Mental Disorders (DSM-5)
* Free from acute exacerbation of their psychosis for at least 3 months prior to Screening
* Clinical Global Impression - Severity (CGI-S) score ≤ 4
* Body mass index (BMI) within 2 standard deviations of, age- and gender-specific body measurements (based on CDC Clinical Growth Chart, 2000)
* Ability to swallow capsules

Main Exclusion Criteria:

* Has a primary psychiatric diagnosis other than schizophrenia or schizoaffective disorder
* Reports having experienced suicidal ideation within 6 months prior to Screening, any suicidal behavior within 2 years prior to Screening based on the Columbia-Suicide Severity Rating Scale (C-SSRS), and/or the investigator assesses the patient to be a safety risk to him/herself or others
* Clinically significant abnormality within 2 years of Screening that in the Investigator's opinion may place the patient at risk or interfere with study outcome variables
* History of a clinically significant cardiac disorder and/or abnormal screening electrocardiogram (ECG) or a QT interval corrected for heart rate using Fridericia formula > 450 msec in males or > 470 msec in females

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2021-03-12 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Site, Principal Investigator — Atlanta, Georgia, United States, 30331; Clinical Site, Principal Investigator — Decatur, Georgia, United States, 30030; Clinical Site, Principal Investigator — Hollywood, Florida, United States, 33024
Locations (3):
- United States (3):
  - Clinical Site, Hollywood, Florida
  - Clinical Site, Atlanta, Georgia
  - Clinical Site, Decatur, Georgia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Lumateperone 42 mg once daily was evaluated in the study. Lumateperone 28 mg once daily was a potential dosage, however it was not evaluated in the study.
Period: Overall Study
Arm/Group | Lumateperone 42 mg Once Daily for 5 Days
Started | 26
Completed | 21
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | Lumateperone 42 mg Once Daily for 5 Days
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.2 (1.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 26
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 26
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics: Cmax
Description: Maximum plasma concentration of lumateperone
Time Frame: Day 1 and Day 5
Population: The PK Analysis Population included all patients who received at least one dose of study drug, had no major protocol deviation that may have impacted PK analyses, and had measurable plasma concentrations to provide an estimate of at least Cmax or AUC.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Lumateperone 42 mg Once Daily for 5 Days
Number analyzed (Participants) | 25
ng/mL
  Day 1 | 19.12 (11.21)
  Day 5: number analyzed (Participants) | 20
  Day 5 | 23.22 (12.60)

2. Primary Outcome: Pharmacokinetics: Tmax
Description: Time of maximum concentration of lumateperone in plasma
Time Frame: Day 1 and Day 5
Population: as for outcome 1
Measure: Median (Full Range); unit: h
Arm/Group | Lumateperone 42 mg Once Daily for 5 Days
Number analyzed (Participants) | 25
h
  Day 1 | 1.000 [0.25 to 6.00]
  Day 5: number analyzed (Participants) | 20
  Day 5 | 1.000 [0.50 to 4.00]

3. Primary Outcome: Pharmacokinetics: AUC0-t
Description: Area under the plasma concentration time curve from time zero to the last measurable of concentration of lumateperone
Time Frame: 0 to 24 hours post-dose on Day 1 and Day 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Lumateperone 42 mg Once Daily for 5 Days
Number analyzed (Participants) | 25
h*ng/mL
  Day 1 | 43.612 (21.404)
  Day 5: number analyzed (Participants) | 20
  Day 5 | 54.975 (26.992)

4. Primary Outcome: Pharmacokinetics: AUC0-tau
Description: Area under the plasma lumateperone concentration time curve from time zero to the end of dosing (tau)
Time Frame: 0 to 24 hours post-dose on Day 1 and Day 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Lumateperone 42 mg Once Daily for 5 Days
Number analyzed (Participants) | 22
h*ng/mL
  Day 1 | 48.158 (20.899)
  Day 5: number analyzed (Participants) | 20
  Day 5 | 58.437 (27.792)

5. Primary Outcome: Pharmacokinetics: t1/2
Description: Terminal elimination half-life of lumateperone
Time Frame: Day 1 and Day 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Lumateperone 42 mg Once Daily for 5 Days
Number analyzed (Participants) | 21
h
  Day 1 | 2.208 (0.6162)
  Day 5: number analyzed (Participants) | 18
  Day 5 | 2.681 (1.092)

6. Primary Outcome: Pharmacokinetics: CL/F
Description: Apparent oral clearance of lumateperone
Time Frame: Day 1 and Day 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Lumateperone 42 mg Once Daily for 5 Days
Number analyzed (Participants) | 20
L/h
  Day 1 | 3062.0 (1292.0)
  Day 5 | 947.14 (595.34)

7. Secondary Outcome: Percentage of Subjects With Treatment-emergent Adverse Events
Time Frame: up to 30 days after last dose, up to a total of 35 days
Population: The Safety analysis population included all patients who took at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Lumateperone 42 mg Once Daily for 5 Days
Number analyzed (Participants) | 26
Participants | 16

8. Secondary Outcome: Change From Baseline in Systolic and Diastolic Blood Pressure
Time Frame: Baseline and Day 6
Population: The Safety analysis population included all patients who took at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Lumateperone 42 mg Once Daily for 5 Days
Number analyzed (Participants) | 21
mmHg
  Supine Systolic Blood Pressure | 0.7 (10.74)
  Diastolic Systolic Blood Pressure | -0.5 (6.64)

9. Secondary Outcome: Change From Baseline in ECG QT Interval
Description: QTcF
Time Frame: Baseline and Day 6
Population: The Safety analysis population included all patients who took at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Lumateperone 42 mg Once Daily for 5 Days
Number analyzed (Participants) | 21
msec | -3.4 (15.19)

10. Secondary Outcome: Change From Baseline in Hemoglobin
Time Frame: Baseline and Day 6
Population: The Safety analysis population included all patients who took at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Lumateperone 42 mg Once Daily for 5 Days
Number analyzed (Participants) | 21
g/dL | -0.50 (0.959)

11. Secondary Outcome: Change From Baseline in White Blood Cell Count
Time Frame: Baseline and Day 6
Population: The Safety analysis population included all patients who took at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: cells*10^9/L
Arm/Group | Lumateperone 42 mg Once Daily for 5 Days
Number analyzed (Participants) | 21
cells*10^9/L | -0.24 (1.173)

12. Secondary Outcome: Change From Baseline in Aspartate Aminotransferase
Time Frame: Baseline and Day 6
Population: The Safety analysis population included all patients who took at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Lumateperone 42 mg Once Daily for 5 Days
Number analyzed (Participants) | 20
U/L | -4.0 (2.78)

13. Secondary Outcome: Change From Baseline in Alanine Aminotransferase
Time Frame: Baseline and Day 6
Population: The Safety analysis population included all patients who took at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Lumateperone 42 mg Once Daily for 5 Days
Number analyzed (Participants) | 20
U/L | -3.2 (2.81)

14. Secondary Outcome: Change From Baseline in Abnormal Involuntary Movement Scale (AIMS)
Description: AIMS is a measure of facial and oral movements, extremity movements and trunk movements. The AIMS total score is reported based on 7 items (items 1 through 7). Each item is rated on a scale from none (0) to severe (4). The AIMS total score ranges from 0 to 28. Higher values of total AIMS score indicate increased severity in abnormal movement.
Time Frame: Baseline and Day 6
Population: The Safety analysis population included all patients who took at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lumateperone 42 mg Once Daily for 5 Days
Number analyzed (Participants) | 21
score on a scale | 0.0 (0.00)

ADVERSE EVENTS:
Time Frame: up to 30 days after last dose, up to a total of 35 days
Arm/Group | Lumateperone 42 mg Once Daily for 5 Days
All-Cause Mortality (participants affected / at risk) | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26
Other Adverse Events (participants affected / at risk) | 16/26
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lumateperone 42 mg Once Daily for 5 Days (N=26)
Nausea (Gastrointestinal disorders) | 7
Vomiting (Gastrointestinal disorders) | 5
Dizziness (Nervous system disorders) | 4
Headache (Nervous system disorders) | 6
Somnolence (Nervous system disorders) | 4
Orthostatic hypotension (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-02-28): https://cdn.clinicaltrials.gov/large-docs/77/NCT04779177/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-09): https://cdn.clinicaltrials.gov/large-docs/77/NCT04779177/SAP_001.pdf